

## NON-INTERVENTIONAL (NI) STUDY PROTOCOL

## **Study information**

| Title | Coronavirus Disease 2019 (COVID-19) Vaccination and Breakthrough Infections Among Persons with Immunocompromising Conditions in the United States |
|---|---|
| Protocol number | C4591035 |
| Protocol version identifier | 1.0 |
| Date | 25 August 2021 |
| EU Post Authorization Study (PAS) register number | Study is not a post-approval safety study (PASS) and is not registered |
| | Date assessed: 09 August 2021 |
| Active substance | Tozinameran |
| Medicinal product | Research name: BNT162b2 |
| | Brand name: Comirnaty |
| Research question and objectives | Primary Objectives |
| Research question and objectives | Primary Objectives Aim 1: Describe profiles, vaccine utilization and resource use among subjects with immunocompromising (IC) conditions vaccinated with BNT162b2 |
| Research question and objectives | Aim 1: Describe profiles, vaccine utilization and resource use among subjects with immunocompromising (IC) conditions |

## Secondary Objectives Evaluate Aims 1, 2, 3 and healthcare resource utilization (HCRU) / costs over time and stratified by relevant patient characteristics (eg, age), in specific IC conditions and by vaccination type (eg, any Messenger ribonucleic acid (mRNA)). **Exploratory Objective** Generate early estimates of the effectiveness of BNT162b2 in preventing COVID-19 infection, stratified by relevant patient characteristics (eg. age) and in specific IC conditions. While the analyses will be focused on the IC population, analyses will also be conducted (in part or entirely) on the non-IC population, the total (IC + non-IC) population or relevant subgroups (eg, other high-risk conditions, vaccination status) to support the interpretation of findings. PPD Author (see section below for full list of study investigators)

This document contains confidential information belonging to Pfizer. Except as otherwise agreed to in writing, by accepting or reviewing this document, you agree to hold this information in confidence and not copy or disclose it to others (except where required by applicable law) or use it for unauthorized purposes. In the event of any actual or suspected breach of this obligation, Pfizer must be promptly notified.

# 1. TABLE OF CONTENTS 2. LIST OF ABBREVIATIONS ......5 6. RATIONALE AND BACKGROUND......9 7. RESEARCH QUESTION AND OBJECTIVES ......10 8. RESEARCH METHODS ......11 8.2.1. Inclusion criteria 12 8.4. Data sources 21 8.6. Data management 22 9. PROTECTION OF HUMAN SUBJECTS .......25 9.1. Patient information. 9.2. Patient consent. 25 9.3. Institutional review board (IRB)/Independent ethics committee (IEC)......25 10. MANAGEMENT AND REPORTING OF ADVERSE EVENTS/ADVERSE 11. PLANS FOR DISSEMINATING AND COMMUNICATING STUDY RESULTS.......26 12. REFERENCES 27

### BNT162b2 C4591035 NON-INTERVENTIONAL STUDY PROTOCOL v1.0, 25 August 2021

| ANNEX 1. LIST OF STAND ALONE DOCUMENTS | 31 |
|-----------------------------------------------|----|
| ANNEX 2. ENCEPP CHECKLIST FOR STUDY PROTOCOLS | 31 |
| ANNEX 3. ICD-10 CODE LIST | 31 |

## 2. LIST OF ABBREVIATIONS

| Abbreviation | Definition |
|--------------|-------------------------------------------------------|
| ACE | Angiotensin Converting Enzyme Inhibitors |
| AIDS | Acquired Immunodeficiency Syndrome |
| ARB | Angiotensin-Receptor Blockers |
| CDC | Centers for Disease Control and Prevention |
| CDM | Charge Description Master |
| CI | Confidence Interval |
| CKD | Chronic Kidney Disease |
| CNS | Central Nervous System |
| COVID-19 | Coronavirus Disease 2019 |
| CPT-4 | Current Procedural Terminology, 4th Edition |
| ЕСМО | Extracorporeal Membrane Oxygenation |
| ED | Emergency Department |
| ENCEPP | European Network of Centres for |
| | Pharmacoepidemiology and Pharmacovigilance |
| ESRDEUA | Emergency Use Authorization |
| FDA | US Food and Drug Administration |
| GPP | Guidelines for Good Pharmacoepidemiology<br>Practices |
| HCPCS | Healthcare Common Procedure Coding System |
| HCRU | Healthcare Resource Utilization |
| HIPAA | Health Insurance Portability and Accountability Act |

| HIV | Human Immunodeficiency Virus |
|---|---|
| IC | Immunocompromising |
| ICD | International Classification of Diseases |
| ICD-10-CM | International Classification of Diseases, 10 <sup>th</sup><br>Revision, Clinical Modification |
| ICD-10-PCS | International Classification of Diseases, 10 <sup>th</sup><br>Revision, Procedure Coding System |
| ICU | Intensive Care Unit |
| IEC | Independent Ethics Committee |
| IgA | Immunoglobulin A |
| IgG | Immunoglobulin G |
| IM | Immuno-Modulators |
| IMV | Invasive Mechanical Ventilation |
| IRB | Institutional Review Board |
| IS | Immunosuppressive |
| ISPE | International Society for Pharmacoepidemiology |
| J&J | Johnson & Johnson |
| LOS | Length of Stay |
| mRNA | Messenger Ribonucleic Acid |
| N | Number |
| N/A | Not Applicable |
| NDC | National Drug Code |
| NEC | Not Elsewhere Classified |
| NOS | Not Otherwise Specified |

| PASS | Post-Approval Safety Study |
|---|---|
| PCS | Procedure Coding System |
| PCV | Proportion of Subjects with Breakthrough SARS-<br>CoV-2 Infections that are Vaccinated |
| PV | Proportion of the Population that is Vaccinated |
| Q1 | First Quartile |
| Q3 | Third Quartile |
| QC | Quality Check |
| RCT | Randomized Controlled Trial |
| RTIE | Real-Time Insights and Evidence |
| SARS-CoV-2 | Severe Acute Respiratory Syndrome Coronavirus 2 |
| SD | Standard Deviation |
| STROBE | Strengthening the Reporting of Observational<br>Studies in Epidemiology |
| US | United States |
| VE | Vaccine Effectiveness |
| Vx | Vaccine |
| WBCs | White Blood Cells |
| WHO | World Health Organization |

## 3. RESPONSIBLE PARTIES

## Principal Investigator(s) of the Protocol

| Name | Job Title | Affiliation / Email | Address |
|------|-----------|------------------------|---------------------------------|
| PPD | PPD | Pfizer / PPD | Pfizer,<br>Collegeville |
| PPD | PPD | Pfizer / PPD | Pfizer, NYC |
| PPD | PPD | Genesis Research / PPD | Genesis<br>Research,<br>Hoboken |
| PPD | PPD | Pfizer / PPD | Pfizer, Madrid |
| PPD | PPD | PPD | Pfizer,<br>Collegeville |
| PPD | PPD | Pfizer / PPD | Pfizer, NYC |
| PPD | PPD | Pfizer / PPD | Pfizer,<br>Collegeville |
| PPD | PPD | Pfizer / PPD | Pfizer, NYC |
| PP D | PPD | Pfizer / PPD | Pfizer,<br>Collegeville |
| PPD | PPD | Pfizer / PPD | Pfizer, NYC |
| PPD | PPD | Pfizer / PPD | Pfizer,<br>Collegeville |
| PPD | PPD | Pfizer / PPD | Pfizer, NYC |

## 4. AMENDMENTS AND UPDATES

None.

#### 5. MILESTONES

| Planned date |
|------------------------------------------------------|
| 09 August 2021 |
| 20 August 2021 |
| 09 August 2021 – 24 August 2021 |
| 25 August 2021 (anticipated) |
| 30 December 2021 |
| Interim: 23 September 2021<br>Final: 28 January 2022 |

#### 6. RATIONALE AND BACKGROUND

In December of 2019, the first cluster of cases of coronavirus disease 2019 (COVID-19), caused by severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection, were reported to the World Health Organization. By the end of 2020, the number of COVID-19 cases in the United States had reached 20,402,814 with 369,742 deaths attributed to the illness. In December 2020 two vaccines were issued Emergency Use Authorization (EUA) by the United States (US) Food and Drug Administration (FDA) for active immunization to prevent COVID-19: BNT162b2 (Pfizer/BioNTech) and mRNA1273 (Moderna). A third vaccine (Ad26.COV2.S, Janssen) was issued EUA on 27 February 2021. These three vaccines demonstrated efficacy in randomized controlled trials (RCTs) against COVID-19 illness, including severe disease; the mRNA vaccines demonstrated efficacies of 94% to 95% in preventing symptomatic COVID-19 illness. At the time of this study, the mRNA vaccines were the most widely administered in the US and evidence is accumulating under real-world conditions that they are highly effective for protecting against SARS-CoV-2 infection, symptomatic COVID-19 illness, and COVID-19-related hospitalization and death, with findings generally consistent with the RCTs.

As vaccination coverage continues to increase across the US and in other countries, it is important to understand vaccine effectiveness (VE) in subpopulations, especially those who were under-represented in RCTs, may have suboptimal immune responses to vaccines, and may be at higher risk for COVID-19-related complications, such as those persons with an immunocompromising (IC) condition. There is emerging real-world evidence that people with an IC condition may not develop as a robust of an immune response as the general population to COVID-19 vaccines and are at increased risk of poor outcomes. Currently, there is sparse information in the published literature on whether suboptimal generation of an

immune response to the COVID-19 mRNA vaccines in people with an IC condition leads to reduced VE. In the RCTs of the mRNA vaccines, those with an IC condition were largely excluded from the study populations. <sup>13, 14</sup> A few recently conducted real-world studies that contained subpopulations with IC conditions have found that while the COVID-19 vaccines were effective in this patient group, VE against SARS-CoV-2 infection, symptomatic illness, and COVID-19-related hospitalization was lower than observed in the general populations of these studies. <sup>15-23</sup>

On 12 August 2021, the FDA amended the EUA for the mRNA COVID-19 vaccines to allow for the use of an additional dose for certain immunocompromised subjects with moderate to severe IC conditions. According to the Centers for Disease Control and Prevention (CDC) guidelines (COVID-19 Vaccines for Moderately to Severely Immunocompromised People | CDC), the additional dose should be administered at least 28 days following the two-dose regimen of the same vaccine to individuals 18 years of age or older (ages 12 or older for Pfizer-BioNTech) who have undergone solid organ transplantation, or who are diagnosed with conditions that are considered to have an equivalent level of immunocompromise. A third dose of the same Mrna vaccine should be used; however, if the Mrna vaccine product given for the first two doses is not available or is unknown, either Mrna COVID-19 vaccine product may be administered.

Further study of patients with various IC conditions is warranted to gain a better understanding of which IC conditions may predispose people to reduced COVID-19 VE to guide further prevention efforts.

#### 7. RESEARCH QUESTION AND OBJECTIVES

The overall objective of this study is to evaluate characteristics, vaccine utilization and outcomes among vaccinated subjects with IC conditions. The primary analysis will be conducted on subjects vaccinated with BNT162b2. A variety of subgroup analyses are planned, along with multiple sensitivity analyses that will test how variations in study design affect results.

#### **Primary Objectives:**

- **Aim 1:** Describe profiles, vaccine utilization and resource use among subjects with IC conditions vaccinated with BNT162b2
- **Aim 2:** Evaluate incidence rates of breakthrough infections among subjects with IC conditions fully vaccinated with BNT162b2
- **Aim 3**: Evaluate the clinical presentation of vaccine breakthrough cases among subjects with IC conditions, including time to infection and severity of disease (hospitalization, mortality)

#### **Secondary Objectives**

Evaluate Aims 1, 2, 3 and HCRU/costs over time and stratified by relevant patient characteristics (eg, age), in specific IC conditions and by vaccination type (eg, any Mrna).

#### **Exploratory Objective**

Generate early estimates of the effectiveness of BNT162b2 in preventing COVID-19 infection, stratified by relevant patient characteristics (eg, age), in specific IC conditions.

#### 8. RESEARCH METHODS

#### 8.1. Study design

This study will be a retrospective database analysis utilizing data sets within the HealthVerity database (Philadelphia, Pennsylvania) covering the time period 01 December 2018 through 08 July 2021 (or latest data available) to describe the characteristics of subjects with IC conditions vaccinated with BNT162b2 and to evaluate the incidence of SARS-CoV-2 breakthrough infections.

Study period: 01 December 2018 – 08 July 2021 (or latest data available)

Index identification period: 11 December 2020 – 08 July 2021 (or latest data available; inclusive)

Index date: The first record for a SARS-CoV-2 vaccine (primary analysis: BNT162b2; sensitivity analyses: any Mrna, any authorized vaccine) from a medical claim, pharmacy claim, or chargemaster record.

Baseline period: 12-month period prior to the index vaccination date

Follow-up period: Variable period beginning after the index date and continuing until the earliest of the following: end of the study or end of continuous insurance enrollment.

#### 8.2. Setting

The primary analysis of this study will include all people at least 12 years of age with at least one vaccine claim (primary analysis: BNT162b2; sensitivity analyses: any Mrna, any authorized vaccine) between 11 December 2020 and 08 July 2021 (or latest date available) from the HealthVerity HealthCare Database. Patients included in the study will be required to have 12 months of continuous medical enrollment prior to the receipt of their first vaccine and have no evidence of a SARS-CoV-2 infection in the year prior to being vaccinated.

The study population will be stratified into two cohorts: non-immunocompromised and immunocompromised. Patients with IC conditions will be identified using a modified implementation of an algorithm developed by Greenberg et al – and later modified and

expanded by Patel et al – for administrative claims based on claims and healthcare records identified in the 12 month baseline period. 24, 25

#### 8.2.1. Inclusion criteria

Patients must meet all of the following inclusion criteria to be eligible for inclusion in the study:

- 1. Unique enrollees in the HealthVerity Vaccine dataset any time after 10 December 2020
- 2. At least 12 years on the index date (ie, first vaccination date)
- No evidence of prior COVID-19 infection (a medical claim, pharmacy claim, or chargemaster record with an International Classification of Diseases, 10<sup>th</sup> Revision, Clinical Modification (ICD-10-CM) diagnosis code of U07.1) in the 12 months prior to the index date
- 4. Have 12 months of continuous enrollment with medical benefits (with or without pharmacy benefits) prior to the index date

Subjects with an IC condition were identified via an algorithm originally developed and validated by Greenberg et al<sup>24</sup> for use in administrative claims database studies. For this study, this algorithm will be modified and expanded based on expert medical opinion. The algorithm is depicted in Figure 1.

Subjects will be identified as immunocompromised if they had ≥1 hospitalization or ≥2 outpatient visits on separate dates with an ICD-10-CM code on a healthcare claim indicating an IC condition or if they had usage of specific immunosuppressive medications during the 12-month baseline period. The IC case definition will incorporate 8 groups based on clinical diagnoses only, 1 group based on both clinical diagnoses and usage of immunosuppressive medication, and 2 other groups based on usage of immunosuppressive medication only, for a total of 11 groups with an IC condition (Figure 1). Subjects with >1 IC condition will also be assessed, for a total of 12 mutually exclusive groups for inclusion in this study. The list of ICD-10-CM codes used to identify IC cases by diagnosis and list of immunosuppressive medications are shown in the Annex

Eight of the disease groups will include subjects with 1) symptomatic human immunodeficiency virus (HIV)/acquired immunodeficiency syndrome (AIDS); 2) solid malignancy; 3) bone marrow transplant; 4) organ transplant (excluding bone marrow); 5) rheumatologic or other inflammatory condition; 6) a primary immunodeficiency; 7) other immune conditions; and 8) chronic kidney disease (CKD) or end stage renal disease (ESRD). Subjects in these IC groups (shown as "Group 1" in Figure 1) will be further stratified by treatment status: those with usage of immunosuppressive medications for >14 days anytime during the baseline period and those without any evidence of >14 days of usage of an immunosuppressive medication during the baseline period. Subjects with a bone marrow or

organ transplant will be further stratified by those who received their 1<sup>st</sup> vaccine dose >100 days prior to their transplant and those who received it <100 days prior to their transplant. Subjects with a solid malignancy will be further stratified by their treatment type: chemotherapy or radiation therapy or immunomodulator, or a mix of these treatments.

The 9<sup>th</sup> subject group (shown as "Group 2" in Figure 1) will include those with a hematologic malignancy, required to have usage of an immunosuppressive medication (chemotherapeutic agent, immunomodulator, or systemic corticosteroid) for >14 days anytime during the baseline period; this subject group will be further stratified by their use of an immunosuppressive medication >6 months or  $\leq$  6 months prior to their index date.

The 10<sup>th</sup> subject group will include subjects with usage of an immunosuppressive medication (chemotherapeutic agent, immunomodulator, or systemic corticosteroid excluding low-dose [<60mg/day] prednisone) for >14 days anytime during the baseline period, but without any ICD-10-CM diagnosis codes indicating the above listed IC conditions on a healthcare claim anytime during the baseline period. Subjects with >14 days usage of antimetabolites anytime during the baseline period will be excluded from this subject group and placed in the 11<sup>th</sup> subject group.

This algorithm differs from that used in Greenberg et al<sup>26</sup> by the following modifications. considered relevant for COVID-19 based on expert medical opinion: the inclusion of subjects with a solid malignancy who had radiation therapy or any treatment mix; the separation of subjects with a bone marrow transplant and those with an organ transplant; the inclusion of chronic inflammatory demyelinating polyneuropathy and immune thrombocytopenic purpura in the "rheumatologic or other inflammatory condition" group; the inclusion of sickle cell disease, asplenia, and psoriatic arthritis in the "other immune disorders" group; the addition of subjects with primary immunodeficiencies and those with CKD or ESRD; the requirement that subjects with a hematologic malignancy have evidence of usage of an immunosuppressive medication; the reclassification of subjects with only usage of an immunosuppressive medication; the removal of subjects with usage of only low dose prednisone; and the inclusion of an ad-hoc group of subjects who had taken anti-metabolites. Additionally, the following subcategories will be created: the first 9 subject groups were stratified according to treatment status; organ transplant subjects will be stratified according to time of receipt of the first COVID-19 vaccine dose in relation to the date of transplant; and subjects with hematologic malignancy will be stratified by time of receipt of treatment relative to their 1st vaccine dose.

When categorizing subjects with the different types of IC conditions, all the subject groups will be mutually exclusive. Subjects meeting the criteria for classification into only a single IC group will be classified accordingly into subject groups 1-11. Any subjects meeting the criteria for classification into multiple IC groups will be categorized into the >1 IC condition group (12<sup>th</sup> subject group).

All subjects will be grouped into an overall study population consisting of subjects identified as having an IC condition or not (i.e., non-IC). Subjects with an IC condition will be further categorized into the specific IC condition groups.

Figure 1: Algorithm to define immunocompromising conditions

Algorithm for case definitions of IC conditions in HealthVerity US claims database



#### 8.3. Variables

Table 1. Immunocompromising Conditions definition

| Variable | Role | Data source(s) | Operational definition |
|---|---|---|---|
| Immunocompromisin<br>g Conditions | Cohort Definition | HealthVerity Vaccine<br>Data | Subjects will be categorized into the following 12 mutually exclusive IC groups based on the algorithm detailed in Figure 1: Symptomatic HIV/AIDs, solid malignancy, bone marrow transplant recipients, organ transplant recipients, rheumatologic or other inflammatory conditions, primary immunodeficiencies, other intrinsic immune conditions, chronic kidney disease or end stage renal disease, hematologic malignancy, immunosuppressive treatment only, antimetabolites only, or >1 IC condition. |

Table 1. Immunocompromising Conditions definition

| Variable | Role | Data source(s) | Operational definition |
|---|---|---|---|
| | | | Subjects falling into more than one of these categories will be categorized as having >1 IC condition. |
| | | | At a minimum, subjects will be required to have one inpatient claim or two outpatient claims on separate days with the IC condition of interest in the baseline period. In cases when >14 days of treatment are required it will be based on the dispensed day supply or distinct days of treatment in the baseline period. |
| | | | The main diagnosis codes to identify IC conditions are presented in ANNEX 1. LIST OF STAND ALONE DOCUMENTS. |

Table 2. Vaccination Status definitions

| Variable | Role | Data source(s) | Operational definition |
|---|---|---|---|
| Any vaccination | Cohort Definition | HealthVerity Vaccine<br>Data | Patients with a claim for any vaccine will be considered vaccinated with any vaccine based on the following codes: |
| | | | Pfizer/BioNTech: 91300, 0001A, 0002A, 59267100001, 59267100002, 59267100003 |
| | | | Moderna: 91301, 0011A, 0012A, 80777027310,80777027399,80777027315, 80777027398 |
| | | | Johnson & Johnson: 91303, 0031A,<br>59676058005,59676058015 |
| | | | Source:<br>https://www.cdc.gov/vaccines/programs/iis/C<br>OVID-19-related-codes html |
| Fully Vaccinated | Cohort Definition | HealthVerity Vaccine<br>Data | Patients will be considered fully vaccinated if they meet any of the following definitions: |
| | | | Two claims for Pfizer/BioNTech vaccine on separate days with >14 days of follow-up after the 2 <sup>nd</sup> vaccination date. No claims for any other vaccines are allowed. |

**Table 2.** Vaccination Status definitions

| Variable | Role | Data source(s) | Operational definition |
|---|---|---|---|
| | | | <ul> <li>Two claims for Moderna vaccine on separate days with &gt;14 days of follow-up after the 2<sup>nd</sup> vaccination date. No claims for any other vaccines are allowed.</li> <li>One claim for the Johnson &amp; Johnson (J&amp;J) vaccine with &gt;14 days of follow-up after the 1<sup>st</sup> vaccination date. No claims for any other vaccines are allowed</li> </ul> |
| Partially vaccinated | Cohort Definition | HealthVerity Vaccine<br>Data | Patients will be considered partially vaccinated if they meet any of the following criteria: • One claim for Pfizer/BioNTech vaccine with > 18 days of follow-up following first vaccination date and no claims for any other vaccine. • One claim for Moderna vaccine with > 25 days of follow-up following first vaccination date and no claims for any other vaccine. • One claim for J&J vaccine with ≤14 days of follow-up following first vaccination date and no claims for any other vaccine. |

Table 3. Patient Characteristics and Vaccine Utilization variable definitions

| Variable | Role | Data source(s) | Operational definition |
|---|---|---|---|
| Age | Patient<br>Characteristics | HealthVerity Vaccine<br>Data | The number of years between the index date and the patient birth year. If multiple birth years are reported for the same HealthVerity ID, the maximum birthyear will be used. Age will be reported in the following categories: 16 – 17, 18 – 29, 30 – 39, 40 – 49, 50 – 64, 65 – 74, 75 – 84, and 85+. Adolescents age 12-15 will also be reported as data accumulates over monthly data cuts. Continuous statistics including mean, standard deviation (SD), median (Q1-Q3), |

Table 3. Patient Characteristics and Vaccine Utilization variable definitions

| Variable | Role | Data source(s) | Operational definition |
|---|---|---|---|
| | | | minimum, and maximum, will also be summarized. |
| Sex | Patient<br>Characteristics | HealthVerity Vaccine<br>Data | Sex will be reported as Male ('M'), Female ('F'), and Unknown |
| US Geographic<br>Region | Patient<br>Characteristics | HealthVerity Vaccine<br>Data | US geographic region will be derived from<br>the patient state and categorized into the<br>following: |
| | | | Northeast – Connecticut, Maine,<br>Massachusetts, New Hampshire, Rhode<br>Island, Vermont, New Jersey, New York,<br>Pennsylvania |
| | | | Midwest – Indiana, Illinois, Michigan, Ohio,<br>Wisconsin, Iowa, Kansas, Minnesota,<br>Missouri, Nebraska, North Dakota, South<br>Dakota |
| | | | South – Delaware, District of Columbia,<br>Florida, Georgia, Maryland, North Carolina,<br>South Carolina, Virginia, West Virginia,<br>Alabama, Kentucky, Mississippi, Tennessee,<br>Arkansas, Louisiana, Oklahoma, Texas |
| | | | West – Arizona, Colorado, Idaho, New<br>Mexico, Montana, Utah, Nevada, Wyoming,<br>Alaska, California, Hawaii, Oregon,<br>Washington |
| | | | Other - Puerto Rico |
| Payer/insurance<br>coverage on index<br>date | Patient characteristics | HealthVerity Vaccine<br>Data | Payer on index date will be reported as the following categories: Commercial, Medicaid, Medicare, Unknown, or missing. If multiple payers are reported on the index date, those will be captured under an ad-hoc "Multiple" category. |
| Vaccine<br>Administration<br>Setting | Patient characteristics | HealthVerity Vaccine<br>Data | Vaccine administration setting will be determined based on the reported place of service for the claim. Prescription claims will be assumed to have occurred in the Pharmacy setting. The most common settings will be reported. |
| Conditions that place<br>or may place patients<br>at risk of Severe<br>COVID-19 (6 months<br>prior) | Patient<br>Characteristics | HealthVerity Vaccine<br>Data | Baseline comorbid conditions that place or<br>may place patients at risk of Severe COVID-<br>19 infection will be assessed in the 6 months<br>prior to index vaccination. The ICD-10-CM,<br>ICD-10 Procedure Coding System (ICD-10- |

Table 3. Patient Characteristics and Vaccine Utilization variable definitions

| Variable | Role | Data source(s) | Operational definition |
|---|---|---|---|
| | | | PCS), Current Procedural Terminology (CPT-4), and Healthcare Common Procedure Coding System (HCPCS) codes used to identify these conditions are based on the Sentinel COVID-19 Natural History Master Protocol (https://www.sentinelinitiative.org/methods-data-tools/methods/master-protocol-development-covid-19-natural-history) |
| Prevention seeking<br>behavior (at baseline) | Patient<br>Characteristics | HealthVerity Vaccine<br>Data | These variables will be assessed during the 12 month baseline period: |
| | | | Telephone or Telehealth visits defined as a claim with any of the following procedure codes (G2012, G2010, G2061-G2063; 99205-99205, 99212-99215, 99421-99423, 99441-99443, G0425-G0427, G0406-G0408) |
| | | | COVID-19 laboratory tests defined as a claim with any of the following CPT-4 codes (87635, 86318, 86328, 86769, 87426, 86408, 86409, 86413) |
| | | | Flu vaccinations defined as a claim with the following procedure codes (90653-90664, 90666-90668, 90724, 90470, 90672, 90673, 90685-90688) |
| | | | The cumulative proportion of IC and non-IC subjects receiving their first dose of COVID-19 vaccine, by month, starting from December 2020 until most recent data. |
| Acute Respiratory<br>Infection<br>Hospitalization (at<br>baseline) | Patient<br>Characteristics | HealthVerity Vaccine<br>Data | Any inpatient claim that occurs in the 12 month baseline period with a diagnosis of J00–J06, J09–J18, J20–J22 will be reported |
| Follow-up time | Patient<br>Characteristics | HealthVerity Vaccine<br>Data | The number of days between the index date and the earliest of the following: end of the study or end of continuous insurance enrollment |
| IS drugs use | Patient<br>Characteristics | HealthVerity Vaccine<br>Data | The proportion of subjects with IC conditions and usage of IS drugs for >14 days during the baseline period will be reported, as well as use within 14 days and 28 days within receipt of the first vaccine dose. IS drugs exclude low-dose [<60mg/day] prednisone. |

Table 3. Patient Characteristics and Vaccine Utilization variable definitions

| Variable | Role | Data source(s) | Operational definition |
|---|---|---|---|
| COVID-19<br>supportive<br>medication use | Patient<br>Characteristics | HealthVerity Vaccine<br>Data | The use of medications considered supportive for COVID-19 will be assessed in the 12-month baseline period including remdesivir, dexamethasone, doxycycline, norepihephrine, methylprednisolone, lopinavir/ritonavir, eculizumab, sarilumab, tocilizumab, losartan, azithromycin, hydroxychloroquine, siltuximab, colchicine, and convalescent plasma. Codes used to identify these treatments will be based on the Sentinel COVID-19 Natural History Master Protocol |
| Other baseline<br>medication use | Patient<br>Characteristics | HealthVerity Vaccine<br>Data | Medications for pre-existing conditions per<br>the Sentinel COVID-19 Natural History<br>Master Protocol (eg, angiotensin converting<br>enzyme inhibitors (ACE), angiotensin-<br>receptor blockers (ARB)). |
| Vaccine utilization | Patient<br>Characteristics | HealthVerity Vaccine<br>Data | Patterns of uptake. The proportion of IC and non-IC patients who are partially and fully vaccinated with BNT162b2 (or any other vaccines), at different calendar months and follow-up periods (eg, 7 days post dose 2, 14 days post dose 2). Mean, median, minimum, and maximum time between receipt of the first and second dose of BNT162b2 (or any other vaccine) |

Table 4. Breakthrough Cases Definition

| Variable | Role | Data source(s) | Operational definition |
|---|---|---|---|
| Breakthrough SARS-<br>CoV-2 infection | Outcome | HealthVerity Vaccine<br>Data | Among patients who meet the definition of fully vaccinated, a breakthrough SARS-CoV-2 infection will be defined by evidence of a claim with a diagnosis code of U07.1 that occurs >14 days after the second vaccination date. The first claim with a diagnosis of COVID-19 after this time will be used to assess mean and median time from the second dose until the breakthrough case |

Table 5. COVID-19 Healthcare resource use and Costs definitions

| Variable | Role | Data source(s) | Operational definition |
|---|---|---|---|
| Emergency<br>department (ED) visit | Outcome | HealthVerity Vaccine<br>Data | An outpatient claim with a place of service = 23 that occurs after the breakthrough COVID-19 diagnosis date or at the same time/episode of care |
| Outpatient Hospital<br>Visit | Outcome | HealthVerity Vaccine<br>Data | An outpatient claim with a place of service = 22 or 19 or a standard billing code that begins with '13' that occurs after the breakthrough COVID-19 diagnosis date or at the same time/episode of care |
| Other Outpatient<br>Visit (not ED, not<br>hospital-based) | Outcome | HealthVerity Vaccine<br>Data | An outpatient claim that does not meet the definition for an ED visit or Outpatient hospital visit. |
| Hospitalization | Outcome | HealthVerity Vaccine<br>Data | A record from the chargemaster data with encounter type of Inpatient OR a series of claims (separated by no more than 2 days) with a place of service = 21 or standard billing codes that begin with '11' or '12' that occur after the breakthrough COVID-19 diagnosis or at the same time/episode of care 1st admission and readmissions will be differentiated. |
| Intensive Care Unit<br>(ICU) | Outcome | HealthVerity Vaccine<br>Data | A claim with a procedure code indicative of ICU utilization during a hospitalization that occurs after the breakthrough COVID-19 diagnosis or at the same time/episode of care 1st admission and readmissions will be differentiated. |
| Invasive Mechanical Ventilation (IMV) / Extracorporeal Membrane Oxygenation (ECMO) | Outcome | HealthVerity Vaccine<br>Data | A claim with a procedure code indicative of IMV/ECMO utilization during a hospitalization that occurs after the breakthrough COVID-19 diagnosis or at the same time/episode of care Includes both 1st admission and readmissions. |
| Inpatient Death | Outcome | HealthVerity Vaccine<br>Data | Death that occurs on or after the date of the breakthrough COVID-19 diagnosis. The date of death will be assumed to be the same as the date of the last recorded encounter in the database. |

Table 5. COVID-19 Healthcare resource use and Costs definitions

| Variable | Role | Data source(s) | Operational definition |
|---|---|---|---|
| | | | Death information is available from the Charge Description Master (CDM) data and is provided as year-month of death only. Time to death will also be explored. |
| Length of Stay (LOS) | Outcome | HealthVerity Vaccine<br>Data | Length of stay (LOS) associated with<br>different types of hospitalization treatments<br>mentioned above (eg, ICU), applicable for<br>first index hospitalization and/or<br>readmissions. |
| Costs | Outcome | HealthVerity Vaccine<br>Data | Non-zero costs associated with any of the previously listed Outpatient and Inpatient encounters (but death). Charges may be assessed in sensitivity analyses to interpret the cost data. |

#### 8.4. Data sources

The HealthVerity database contains the largest all-payer (commercial, Medicare, and Medicaid) collection of US healthcare administrative data that links patients' journeys across inpatient admissions, outpatient visits, laboratory visits, and pharmacy services, including COVID-19 tests and vaccinations. Electronic medical records, including Veradigm data, are integrated with the administrative claims data from multiple sources to capture a relatively complete summary of patients' clinical history, including comorbid conditions and other risk factors that may predispose individuals to infections and complications, and use of healthcare resources. With monthly updates available, this data source provides a nearly real-time longitudinal view of patients' journeys across multiple sites of care. All data sets contained within the HealthVerity database are secured and encrypted and all patient information is deidentified. Thus, the data source is fully compliant with the Health Insurance Portability and Accountability Act (HIPAA).

#### 8.5. Study size

The sample size for this study is fixed by the duration of the observation window. No formal sample size computation will be performed. All subjects who meet the inclusion/exclusion criteria will be included in the analyses.

Feasibility analyses confirmed the availability of data to identify vaccinated subjects, subjects with underlying IC conditions, and breakthrough infections. The current study is mainly descriptive in nature. For the exploratory aim, the entire source population available in the HealthVerity database will be included in the analysis.

#### 8.6. Data management

This study will use secondary data collected in the HealthVerity Healthcare database, specifically from the Vaccine and Real-Time Insights and Evidence (RTIE) data sets, which are de-identified and HIPAA compliant. The study will utilize a data cut consisting of data from December 1, 2018 through July 8, 2021 (or the most recent data available).

#### 8.7. Data analysis

Data analyses will follow extensive feasibility analyses aimed at determining whether a full study and the assessment of vaccine effectiveness are feasible, as illustrated below:

## Study implementation approach



Characteristics of the IC, non-IC and total population (IC + non-IC) groups will be described. Descriptive statistics for continuous variables will include N (number of patients), mean, median, standard deviation, Q1, Q3, minimum, and maximum. Categorical variables will be described using frequency counts and percentages.

The incidence rate of breakthrough cases of SARS-CoV-2 infection will be determined based on the following:

Among fully vaccinated patients, those who have a claim for COVID-19 (ICD-10-CM: U07.1) that occurs on or after >14 days following their second dose of an mRNA vaccine (or 1<sup>st</sup> dose of Johnson & Johnson) will be considered to have had a breakthrough event. The time from 14 days after the qualifying dose until the breakthrough event will be the person time at risk.

 Among fully vaccinated patients with no evidence of COVID-19 after their qualifying dose, the time from 14 days after the qualifying dose until the end of follow-up will be the person time at risk.

The incidence rate of breakthrough cases of SARS-CoV-2 infection will be calculated as the number of patients who experience the event divided by the observed time at risk, and reported per 100 person years. Poisson 95% confidence intervals will be reported for the incidence rates.

Absolute effect measures such as risk difference between non-IC and IC will be reported. Time period specific effect estimates (eg, at 6 months after vaccination) may be estimated if feasible. The characteristics of the breakthrough infections will be described, including clinical presentation and severity.

The primary analysis will describe results among the non-IC cohort and the IC cohort who are vaccinated with BNT162b2. Subgroup analyses will include results for clinically meaningful subgroups as defined by vaccination type, relevant patient characteristics (eg, age), and each IC condition as listed below:

- HIV/AIDS
- Solid malignancy
- Bone marrow transplant
- Organ transplant (excluding bone marrow)
- Rheumatologic/inflammatory
- Primary Immunodeficiencies
- Other immune condition
- CKD or ESRD
- Hematologic malignancy
- IS drug use: >14 days IS medications (chemotherapy, immuno-modulators (IM), or corticosteroids excluding low-dose [<60mg/day] prednisone See Drug List) and not falling into any of the above 9 condition groups
- >14 days of anti-metabolite use and not falling into any of the above 10 condition or drug use groups
- More than 1 IC condition

Analyses for younger cohorts (eg, 12-15) will also be conducted, as data accumulates.

For the exploratory aim, the Screening Method will be used to calculate VE for the overall study population of subjects with an IC condition and also stratified VE estimates for the different immunocompromised subject groups, with VE also determined for those subjects with >1 IC condition<sup>26</sup>. We will use the proportion of the population that are vaccinated (PV) and the proportion of subjects with breakthrough SARS-CoV-2 infections that are vaccinated (PCV) to calculate VE using the following formula:

$$VE = (PV - PCV)/[PV(1-PCV)]$$

where PV = the proportion of the population that is vaccinated (ie, vaccination coverage) and PCV = the proportion of subjects with breakthrough SARS-CoV-2 infections that are vaccinated.

Additionally, breakthrough incidence rates and VE will be stratified by age at diagnosis (eg, < 65 and  $\ge 65$  years of age at index vaccination).

Sensitivity analyses will be conducted to test the robustness of findings by varying key study design aspects (eg, continuous enrolment, IC case definition) and data analysis techniques. Other statistical techniques (eg, matched analyses, multiple regression, propensity scores) may be applied on an exploratory basis after careful examination of potential confounders (eg, age, time from vaccination). Exploratory analyses related to alternate dosing may also be conducted upon feasibility results, and as recommendations from public health authorities evolve. The analyses (entirely or in part) will be conducted over time and updated on a rolling basis as monthly data cuts become available.

While the analyses will be focused on the IC population, analyses will also be conducted (in part or entirely) on the non-IC population, the total (IC + non-IC) population or relevant subgroups (eg, other high-risk conditions, vaccination status) to support the interpretation of findings.

#### 8.8. Quality control

Data in HealthVerity's COVID Healthcare database are collected weekly in an electronic format. HealthVerity employs its foundational product to match patients between different data sources with high accuracy. However, not all data points are available in every data source and as a result, not all variables in the database are completely populated. In addition, the database contains both pre- and post-adjudicated claims and, based on the data source, adjudication may or may not be captured. To maximize data completeness and uniformity, it may be necessary to exclude certain data sources from the analysis due to differences in data structure and content.

#### 8.9. Limitations of the research methods

There are several limitations associated with this study. The healthcare claims data are

collected for billing purposes and may be subject to misclassification, misdiagnosis, and underreporting. While the sensitivity and specificity of the Greenberg algorithm were 87.4% (95% confidence interval (CI), 80.6-92.5%) and 97.6% (95% CI, 95.0-99.9%), we cannot assess the impact that our modifications had on the accuracy of the algorithm to identify immunocompromised patients. While we used the same codes as Patel<sup>25</sup> for HIV, which included HIV only when symptomatic, we cannot be certain about the degree of immunosuppression among patients who had International Classification of Diseases (ICD) codes for symptomatic HIV/AIDS. Further research leveraging Electronic Health Records/ Lab data is warranted to increase sensitivity of capturing symptomatic HIV cases. Due to irregular capture of COVID-19 vaccinations by insurers these results may only be generalizable to a subset of insured individuals. The HealthVerity Census algorithm which links unique patients across disparate data sources may incorrectly assign the same unique identifier to different people or different identifiers to the same person, though this is expected to have negligible impact on the interpretation of results. Additionally, due to the fact that the Health Verity Data set is comprised of multiple data sources, there may be different levels of missingness for certain variables captured in this analysis.

#### 8.10. Other aspects

Not applicable.

#### 9. PROTECTION OF HUMAN SUBJECTS

#### 9.1. Patient information

This study involves data that exist in anonymized structured format and contain no patient personal information.

#### 9.2. Patient consent

As this study involves anonymized structured data, which according to applicable legal requirements do not contain data subject to privacy laws, obtaining informed consent from patients by Pfizer is not required.

#### 9.3. Institutional review board (IRB)/Independent ethics committee (IEC)

IRB/IEC review is not required.

## 9.4. Ethical conduct of the study

The study will be conducted in accordance with legal and regulatory requirements, as well as with scientific purpose, value and rigor and follow generally accepted research practices described in Guidelines for Good Pharmacoepidemiology Practices (GPP) issued by the International Society for Pharmacoepidemiology (ISPE). This study will follow the Strengthening the Reporting of Observational Studies in Epidemiology (STROBE) reporting guideline

# 10. MANAGEMENT AND REPORTING OF ADVERSE EVENTS/ADVERSE REACTIONS

This study involves data that exist as structured data by the time of study start. In these data sources, individual patient data are not retrieved or validated, and it is not possible to link (i.e., identify a potential association between) a particular product and medical event for any individual. Thus, the minimum criteria for reporting an adverse event (AE) (i.e., identifiable patient, identifiable reporter, a suspect product, and event) cannot be met

#### 11. PLANS FOR DISSEMINATING AND COMMUNICATING STUDY RESULTS

A final study report detailing the final study protocol and the analysis results will be provided when the study is complete.

In the event of any prohibition or restriction imposed (e.g., clinical hold) by an applicable competent authority in any area of the world, or if the investigator is aware of any new information which might influence the evaluation of the benefits and risks of a Pfizer product, Pfizer should be informed immediately.

#### 12. REFERENCES

- World Health Organization. Archived: WHO timeline COVID-19. Available from: https://www.who.int/news/item/27-04-2020-who-timeline---covid-19. Accessed July 8, 2021
- Centers for Disease Control and Prevention. COVID data tracker. Available from: https://covid.cdc.gov/covid-data-tracker/#trends\_dailytrendscases. Accessed July 8, 2021.
- US Food and Drug Administration. Pfizer-BioNTech COVID-19 vaccine. Available from: https://www.fda.gov/emergency-preparedness-and-response/coronavirus-disease-2019-covid-19/pfizer-biontech-covid-19-vaccine. Accessed July 8, 2021.
- US Food and Drug Administration. Moderna COVID-19 vaccine. Available from: https://www.fda.gov/emergency-preparedness-and-response/coronavirus-disease-2019-covid-19/moderna-covid-19-vaccine. Accessed July 8, 2021.
- US Food and Drug Administration. Janssen COVID-19 vaccine. Available from: https://www.fda.gov/emergency-preparedness-and-response/coronavirus-disease-2019-covid-19/janssen-covid-19-vaccine. Accessed July 29, 2021.
- Centers for Disease Control and Prevention. Science brief: COVID-19 vaccines and vaccination. Updated May 27, 2021. Available from: https://www.cdc.gov/coronavirus/2019-ncov/science/science-briefs/fully-vaccinated-people.html. Accessed July 19, 2021.
- Williamson EJ, Walker AJ, Bhaskaran K, et al. Factors Associated with COVID-19related death using OpenSAFELY. Nature. 2020;584:430-436.
- Haidar G, Mellors JW. Improving the outcomes of immunocompromised patients with COVID-19. Clin Infect Dis. 2021; May 5;ciab397. Doi: 10.1093/cid/ciab397. Online ahead of print.
- Boyarsky BJ, Werbel WA, Avery RK, et al. Immunogenicity of a single dose of SARS-CoV-2 messenger RNA vaccine in solid organ transplant recipients. JAMA. 2021;325:1784-1786.
- 10. Yi SG, Knight RJ, Graviss EA, et al. Kidney transplant recipients rarely show an early antibody response following the first COVID-19 vaccine administration. Transplantation 2021;105:e72-e73.

- Agha ME, Blake M, Chilleo C, et al. Suboptimal response to COVID-19 mRNA vaccines in hematologic malignancies patients. medRxiv. 2021; Apr 7;2021.04.06.21254949. doi: 10.1101/2021.04.06.21254949. Preprint.
- 12. Boyarsky BJ, Ruddy JA, Connolly CM, et al. Antibody response to a single dose of SARS-CoV-2 mRNA vaccine in patients with rheumatic and musculoskeletal diseases. Ann Rheum Dis. 2021; Mar 23;annrheumdis-2021-220289. Doi: 10.1136/annrheumdis-2021-220289. Online ahead of print.
- Polack FP, Thomas SJ, Kitchin N, et al. Safety and efficacy of the BNT162b2 mRNA COVID-19 vaccine. N Engl J Med. 2020;383:2603-2615.
- Baden LR, El Sahly HM, Essink B, et al. Efficacy and safety of the mRNA-1273 SARS-CoV-2 vaccine. N Engl J Med. 2021;384:403-416.
- Young-Xu Y, Korves C, Powell EI, et al. Coverage and effectiveness of mRNA SARS-CoV-2 vaccines among United States Veterans. medRxiv. Jun 22, 2021. Doi: 10.1101/2021.06.14.21258906.
- 16. Whitaker HJ, Tsang RSM, Byford R, et al. Pfizer-BioNTech and Oxford AstraZeneca COVID-19 vaccine effectiveness and immune response among individuals in clinical risk groups. Khub.net. Preprint. Posted July 2021.
- 17. Tenforde MW, Patel MM, Ginde AA, et al. Effectiveness of SARS-CoV-2 mRNA vaccines for preventing Covid-19 hospitalizations in the United States. medRxiv. Preprint. Posted July 8, 2021.
- 18. Chodick G, et al. The effectiveness of the two-dose BNT162b2 vaccine: analysis of real-world data. Clin Infect Dis. 2021 May 17; Online ahead of print.
- 19. Kahn N & Mahmud N. Effectiveness of SARS-CoV-2 vaccination in a Veterans Affairs cohort of patients with inflammatory bowel disease with diverse exposure to immunosuppressive medications. Gastroenterology. 2021;S0016-5085(21)03066-3. Online ahead of print.
- 20. Yelin I, et al. Associations of the BNT162b2 COVID-19 vaccine effectiveness with patient age and comorbidities. MedRxiv preprint.
- Dagan N, Barda N, Kepten E, et al. BNT162b2 mRNA Covid-19 vaccine in a nationwide mass vaccination setting. N Engl J Med. 2021;384:1412-1423.

- Barda N, Dagan N, Balicer RD. BNT162b2 mRNA Covid-19 vaccine in a nationwide mass vaccination setting: Reply. N Engl J Med. 2021;384:1970.
- 23. Broh-Nissimov T, Orenbuch-Harroch E, Chowers M, et al. BNT162b2 vaccine breakthrough: clinical characteristics of 152 fully vaccinated hospitalized COVID-19 patients. J Clin Microbiol Infect. 2021;S1198-743x(21)00367-0. Online ahead of print.
- 24. Greenberg JA, Hohmann SF, Hall JB, et al. Validation of a method to identify immunocompromised patients with severe sepsis in administrative databases. Ann Am Thorac Soc. 2016;13:253-258.
- 25. Patel M, Chen J, Kim S, et al. Analysis of MarketScan Data for Immunosuppressive Conditions and Hospitalizations for Acute Respiratory Illness, United States. Emerging Infectious Diseases. 2020;26(8):1720-1730.
- 26. Remschmidt C. Application of the screening method to monitor influenza vaccine effectiveness among the elderly in Germany. BMC Infectious Diseases (2015) 15:137

## 13. LIST OF TABLES

| Table 1. | Immunocompromising Conditions definition | 14 |
|---|---|---|
| Table 2. | Vaccination Status definitions | 15 |
| Table 3. | Patient Characteristics and Vaccine Utilization variable definitions | 16 |
| Table 4. | Breakthrough Cases Definition. | 19 |
| Table 5. | COVID-19 Healthcare resource use and Costs definitions | 20 |
| 14. LIST OF 1 | FIGURES | |
| Figure 1: Algo | rithm to define immunocompromising conditions | 14 |

## ANNEX 1. LIST OF STAND ALONE DOCUMENTS

None

## ANNEX 2. ENCEPP CHECKLIST FOR STUDY PROTOCOLS

N/A

#### ANNEX 3. ICD-10 CODE LIST

| IC Condition | ICD-10 Code |
|---|---|
| HIV/AIDS* | B20-B24 |
| Solid malignancy | |
| Organ/system malignant tumors | C00-C07; C11-C19; C22-C80; Z85 |
| Neuroendocrine tumors | C7A; C7B; D3A |
| Neoplasms of uncertain behavior | D00-D49 |
| Bone marrow transplant | Z94.81 |
| Organ transplant | |
| Complications of transplanted organ | T86 |
| Organ transplant status | Z94 except Z94.81; Z98.85 |
| Rheumatologic or other inflammatory condition | |
| Sarcoidosis | D86 |
| Amyloidosis Not Otherwise Specified (NOS) | E85 |
| Familial Mediterranean fever | E85.0; M04 |
| Amyloidosis Not Elsewhere Classified (NEC) | E85.1; E85.3; E85.8 |
| Multiple sclerosis | G35 |
| Other Central Nervous System (CNS) demyelination | G36; G37.1; G37.3; G37.8; G37.9 |
| Acute infective polyneuritis | G61.0; G61.9 |
| Acute myocarditis | I40 |
| Polyarteritis nodosa and other | M30 |
| Allergic alveolitis/pneumonitis NOS | T78.40; J67.9 |
| Other alveolar pneumonopathy | J84.01; J84.02; J84.09 |

| IC Condition | ICD-10 Code |
|---|---|
| Enteritis and colitis | K50-K52 |
| Lupus erythematosus | L93.0; L93.2; M32 |
| Diffuse connective tissue disease | L94; M35.8; M35.9 |
| Arthropathy with infection | M12.9; M01.X0; M02.10 |
| Crystal arthropathies | M11 |
| Rheumatoid arthritis/inflammatory polyarthropathy | M05-M14 |
| Inflammatory spondylopathies | M46 |
| Polymyalgia rheumatica | M31.5; M35.3 |
| Chronic inflammatory demyelinating polyneuropathy | G61.81 |
| Immune thrombocytopenic purpura | D69.3 |
| Primary Immunodeficiency | |
| X-linked agammaglobulinemia | D80.8 |
| Common variable immunodeficiency | D83.1; D83.2; D83.8; D83.9 |
| Immunoglobulin A (IgA) deficiency | D80.2 |
| Immunoglobulin G (IgG) sub-class deficiency | D80.3 |
| Severe combined immunodeficiency | D81.1 |
| Di George syndrome | D82.1 |
| Wiskott-Aldrich | D82.0 |
| Ataxia telangiectasia | G11.3 |
| Interferon-gamma/Interleukin 12 axis deficiencies | D84.89 |
| Persistent complement, properdin or Factor B deficiency | D84.1 |
| Received eculizumab for >14 days in the baseline period | |
| Chronic granulomatous disease | D71 |
| Chediak-Higashi | E70.330 |
| Leukocyte adhesion deficiency | D72: Genetic anomalies of leukocytes |
| Myeloperoxidase deficiency | D72.89: Other specific disorders of White<br>Blood Cells (WBCs) |

| IC Condition | ICD-10 Code |
|---|---|
| Other immune conditions | |
| Disorders of immune mechanism | D89 |
| Neutropenia | D70 |
| Functional disorders of neutrophils | D71 |
| Genetic anomalies of leukocytes | D72.0 |
| Decreased leukocyte count | D72.81 |
| Leukocyte disease NEC | D72.89 |
| Leukocyte disease NOS | D72.9 |
| Myelofibrosis | D75.81 |
| Blood diseases NEC | D47.4; D75.89; D75.9; D89.2 |
| Blood diseases NOS | D75.9; D75.89 |
| Immunologic findings NEC | R76; R83.4-R87.4; R89.4 |
| Nonspecific immune findings NEC and NOS | R76; R83.4-R87.4; R89.4 |
| Sickle cell disease | D57 |
| Asplenia | Q89.01 |
| Psoriatic arthritis | L40.52 |
| Kidney condition | |
| Chronic kidney disease | A18.11; A52.75; B52.0; C64.x; C68.9; D30.0x; D41.0x-D41.2x; D59.3; E08.2x; E09.2x; E10.2x; E10.65; E11.2x; E11.65; E13.2x; E74.8; I12.xx; I13.0; I13.1x; I13.2; K76.7; M10.3x; M32.14; M32.15; N01.x-N08.x; N13.1; N13.1x-N13.39; N14.x; N15.0; N15.8; N15.9; N16; N17.x; N18.1-N18.5; N18.8; N18.9; N19; N25.xx; N26.1; N26.9; O10.4xx; O12.xx; O26.83x; O90.89; Q61.02; Q61.1x-Q61.8; Q26.0-Q26.39; R94.4 |
| End stage renal disease | N18.6 AND on dialysis (any type): Z99.2;<br>Z49; Z9115; Z4931; OR Z4901 |
| On hemodialysis | Any subject with the ESRD codes above and ≥1 hemodialysis procedure session during the baseline period identified by at ≥1 of the following codes: Z49.31; |

| IC Condition | ICD-10 Code |
|---|---|
| | Z49.32; I953; A4680; A4690; A4706-<br>A4709; A4730; A4740; A4750; A4755;<br>A4802; A4870; A4890; A4918; E1520;<br>E1530; E1540; E1550; E1560; E1575;<br>E1580; E1590; E1600; E1610; E1615;<br>E1620; E1625; E1636; G0365; G0392;<br>G0393; G8081; G8082; G8085; S9335;<br>90935; 90937; 90940; 93990; 36800;<br>36810; 36815 |
| On peritoneal dialysis | Any subject with the ESRD codes above and ≥1 peritoneal dialysis procedure session during the baseline period identified by ≥1 of the following codes: Z49.02; 90945; 90947 |
| Hematologic malignancy** | |
| Lymphatic and hematopoietic tissue malignancy | C81-C83; C88-C96 |

CNS: central nervous system; ICD-10: International Classification of Diseases, 10th Revision; IgG: Immunoglobulin G, IgA: Immunoglobulin A, NOS: not otherwise specified; NEC: necrotizing enterocolitis; WBCs: White blood cells.

<sup>\*</sup>Excluded asymptomatic HIV code of ICD-10: Z21.

<sup>\*\*</sup>Required to have usage of an immunosuppressive medication (chemotherapeutic agent, immunomodulator, or systemic corticosteroids) for >14 days anytime during the baseline period.